CLINICAL TRIAL: NCT01810965
Title: Impact of Bloodletting on Iron Metabolism in Type 1 Hemochromatosis: Pathophysiological and Clinical Implications. Pilot Study.
Brief Title: Impact of Bloodletting on Iron Metabolism in Type 1 Hemochromatosis
Acronym: SAIFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANSM 2012-A01392-41
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Hemochromatosis Type 1
Keywords: Hemochromatosis type 1
MeSH Terms: conditions — Hemochromatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort (Experimental)
  Interventions: Procedure: First evaluation phase : no intervention / Second evaluation phase: bloodletting of 7 ml/kg (with a maximum of 500ml)

INTERVENTIONS:
Procedure: First evaluation phase : no intervention / Second evaluation phase: bloodletting of 7 ml/kg (with a maximum of 500ml)

SUMMARY:
Hemochromatosis type 1 is one of the most frequent genetic disease since the genetic predisposition (homozygosity for the C282Y mutation of the HFE gene) is encountered in about 3/1000 white subjects (5/1000 in Brittany, France).

For the half of these predisposed subjects, the phenotypic expression of the disease needs a treatment. This treatment is based upon repeated bloodletting which is generally considered as simple, safe and effective.

Nevertheless, it is still questioned as regard its physiopathological justification and its clinical implications. Indeed, bloodletting could cause an increase of non-transferrin bound iron (NTBI) particularly for its reactive form called labile plasma iron (LPI) This adverse physiopathological effect could have clinical consequences and could be linked with articular consequences which can be aggravated by the treatment.

DETAILED DESCRIPTION:
Hemochromatosis type 1 is one of the most frequent genetic disease since the genetic predisposition (homozygosity for the C282Y mutation of the HFE gene) is encountered in about 3/1000 white subjects (5/1000 in Brittany, France).

For the half of these predisposed subjects, the phenotypic expression of the disease needs a treatment. This treatment is based upon repeated bloodletting which is generally considered as simple, safe and effective.

Nevertheless, it is still questioned as regard its physiopathological justification and its clinical implications. Indeed, bloodletting could cause an increase of non-transferrin bound iron (NTBI) particularly for its reactive form called labile plasma iron (LPI) This adverse physiopathological effect could have clinical consequences and could be linked with articular consequences which can be aggravated by the treatment.

The primary objective is to explore the effect of bloodletting upon plasmatic concentrations of NTBI.

The secondary objectives are to:

* explore the impact of bloodletting upon different parameters of iron metabolism and in particular LPI, hepcidinemia and markers of erythropoiesis ;
* explore basal and nycthemeral characteristics of new parameters of iron metabolism (hepcidin, NTBI, LPI) in hemochromatosis patients.

The demonstration of an adverse effect of bloodletting upon iron metabolism would allow for a therapeutic innovation based upon an association of bloodletting and oral chelation during the induction treatment of type 1 hemochromatosis and, more generally in hepcidino deficient forms of hemochromatosis.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Age 18 years or older
* Homozygosity for the C282Y mutation of the HFE gene
* With an indication of treatment by bloodletting (in accordance with the French HAS guidelines)
* Ferritinemia ≥ 500µg/L
* Transferrin saturation ≥ 75%
* Never treated by bloodletting
* Written informed consent

Exclusion Criteria:

* Contraindication to bloodletting
* Chronic inflammatory or dysmetabolic or neoplastic disease
* Major cardiovascular disease
* Excessive consumption of alcohol (≥ 3gr/day)
* Treatment by iron chelators, C or E vitamins
* Stay in altitude> 1500m in the month preceding the period Day 1
* Patients under guardianship
* Blood donation in the 3 past months
* Night / shift workers

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-06-03 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Maximal variation (delta maximum) of NTBI during the 5 days following a bloodletting | Day 5

SECONDARY OUTCOMES:
Kinetic of NTBI plasmatic concentration during the 5 days following a bloodletting | Day 5
Maximal variation (delta maximum) of LPI during the 5 days following a bloodletting | Day 5
Maximal variation (delta maximum) of hepcidin during the 5 days following a bloodletting | Day 5
Kinetic of LPI plasmatic concentration during the 5 days following a bloodletting | Day 5
Kinetic of hepcidin plasmatic concentration during the 5 days following a bloodletting | Day 5
CRP | Day 9, day 10, day 11 and day 12
Hemoglobin | Day 9, day 10, day 11 and day 12
Soluble transferrin receptor | Day 9, day 10, day 11 and day 12
EPO | Day 9, day 10, day 11 and day 12
Circadian kinetic of NTBI plasmatic concentration when no bloodletting is performed | Day 1
Circadian kinetic of API plasmatic concentration when no bloodletting is performed | Day 1
Circadian kinetic of hepcidine plasmatic concentration when no bloodletting is performed | Day 1
Maximal variation (delta maximum) of transferrin saturation during the 5 days following a bloodletting | Day 5
Kinetic of transferrin saturation during the 5 days following a bloodletting | Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Martine Ropert-Bouchet, MD, Principal Investigator — Rennes University Hospital; Bruno Laviolle, MD, PhD, Study Chair — Rennes University Hospital
Locations (1):
- CHU Pontchaillou, Rennes, France